CLINICAL TRIAL: NCT01264861
Title: Open-Label Escalating Dose Study Using [123|]ß-CIT SPECT Single Photon Emission Computerized Tomography (SPECT) to Evaluate Dopamine and Serotonin Transporter Occupancy by Safinamide in Parkinson Disease Patients
Brief Title: A Study to Evaluate Safinamide's Effect on Dopamine and Serotonin's Availability by Using Brain Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Dopamine transporter brain imaging trial is terminated due to a company decision to return all rights for Safinamide back to Newron Pharmaceuticals
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 28849
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Parkinson Disease
Keywords: Evaluate dopamine and serotonin activity in the brain at 3 doses of Safinamide
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: (Experimental): Arm 1: Eligible subjects will receive escalating doses of safinamide for the 6-week duration of treatment. Each dose level will be last 10-14 days. Doses 200mg and 300mg will have a 3 day intermediate step up dose, 150mg and 250mg dose.
  Interventions: Drug: Safinamide

INTERVENTIONS:
Drug: Safinamide — Safinamide 100 mg/day = two 50 mg tablets administered orally, once a day, in the morning, with or without food.
  Safinamide 200 mg/day = four 50 mg tablets administered orally, once a day, in the morning, with or without food; this will be preceded by a three day titration of 150 mg = three 50 mg tablets administered orally, once a day, in the morning, with or without food.
  Safinamide 300 mg/day = six 50 mg tablets administered orally, once a day, in the morning, with or without food; this will be preceded by a three day titration of 250 mg = five 50 mg tablets administered orally, once a day, in the morning, with or without food.

SUMMARY:
This is a study of safinamide, an investigational drug for Parkinson disease (PD). Safinamide is being developed as add-on therapy for the treatment of Parkinson disease. It is theorized that safinamide acts by increasing the available dopamine in those areas of the brain where dopamine is decreased as a result of Parkinson;s Disease. . Dopamine in the brain is involved in controlling body movements. Safinamide has been extensively studied in animals, and has been shown to increase the level of dopamine in these animals. Safinamide has also been tested in patients with Parkinson disease. The goal of this research trial is to see if safinamide is safe and well tolerated and to better understand how it affects the dopamine system in the brain in individuals with Parkinson disease. Data from this trial may provide essential information about the effectiveness and safety of these doses of safinamide in patients with early Parkinson disease, who are already receiving a stable dose of their normal Parkinson disease treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 40-80 years of age.
2. Subject must have a diagnosis of idiopathic Parkinson's disease, and a Hoehn and Yahr stage of I-III.
3. Subjects must be concomitantly treated with a stable dose of a single dopamine agonist prior to the screening visit.
4. Subjects must be able to understand and willing to sign an approved Informed Consent form.
5. Female subjects must be neither pregnant or breast-feeding.

Exclusion Criteria:

1. Subjects with any form of Parkinsonism other than idiopathic Parkinson's disease.
2. Subjects currently experiencing motor fluctuations (end of dose wearing off), dyskinesias, or significant postural hypotension.
3. Subjects treated with l-dopa, anticholinergics, amantadine, MAO inhibitors, COMT inhibitors, tricyclic antidepressants, and / or SSRI and SNRI antidepressants.
4. Subjects with a history of psychosis, either previously or currently, or a score ≥ 3 on item 2 or 3 of the UPDRS Part I.
5. Subjects with evidence of dementia or cognitive dysfunction.
6. Subjects with current diagnosis of substance abuse or history of alcohol or drug abuse in the past three months.
7. Subjects with current clinically significant gastrointestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease, including hypertension that is not well controlled, asthma, chronic obstructive pulmonary disease, and Type I diabetes.
8. Subjects with a concomitant disease likely to alter absorption, metabolism or elimination of the study drug.
9. Female subjects must be neither pregnant nor lactating.
10. Subjects with hypersensitivity or contraindications to MAO-B inhibitors.
11. Subjects with a neoplastic disorder, which is either currently active or has been in remission for less than one year.
12. Subjects with second- or third-degree atrio-ventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction within three months of the screening visit, or significant ECG abnormality, including QTc ≥ 450 msec (males) or ≥ 470 msec (females), where QTc is based on Bazett's correction method.
13. Subjects with a history or a current diagnosis of human immunodeficiency virus infection, or tests positive for Hepatitis B surface antigen, tests positive for Hepatitis B core antibody, but negative for Hepatitis B surface antibody, or tests positive for Hepatitis C antibodies.
14. Subjects who have participated in a previous clinical trial with safinamide, have participated in a previous clinical trial within 30 days of entry into the study, or have received treatment with any investigational compound within thirty days or five half-lives, whichever is longer, prior to screening.
15. Subjects with any abnormality that the investigator deems to be clinically relevant.
16. Legal incapacity or limited legal capacity
17. Other significant disease that in the Investigator's opinion would exclude the subject from the trial.
18. Treatment with a drug that has hepatotoxic potential within 4 weeks, or received radiation therapy or a drug with cytotoxic potential within one year prior to the screening visit.
19. Ophthalmologic history including any of the following conditions: albino subjects, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity, retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation, or diabetic retinopathy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01-24 (Actual)

PRIMARY OUTCOMES:
The percent change from baseline to steady state (end of dosing period for 100 mg daily safinamide doses) on quantitative determinations of occupancy of the dopamine transporter in striatum as determined by [123|] ß-CIT SPECT scanning. | Every two weeks for six weeks
The percent change from baseline to steady state (end of dosing period for 200 mg daily safinamide doses) on quantitative determinations of occupancy of the dopamine transporter in striatum as determined by [123|] ß-CIT SPECT scanning. | Every two weeks for six weeks
The percent change from baseline to steady state (end of dosing period for 300 mg daily safinamide doses) on quantitative determinations of occupancy of the dopamine transporter in striatum as determined by [123|] ß-CIT SPECT scanning. | Every two weeks for six weeks

SECONDARY OUTCOMES:
The percent change from baseline to steady state (end of dosing period for 100 mg daily safinamide doses) on quantitative determinations of occupancy of the serotonin transporter in brainstem as determined by [123|] ß-CIT SPECT scanning. | Every two weeks for six weeks
The percent change from baseline to steady state (end of dosing period for 200 mg daily safinamide doses) on quantitative determinations of occupancy of the serotonin transporter in brainstem as determined by [123|] ß-CIT SPECT scanning. | Every two weeks for six weeks
The percent change from baseline to steady state (end of dosing period for 300 mg daily safinamide doses) on quantitative determinations of occupancy of the serotonin transporter in brainstem as determined by [123|] ß-CIT SPECT scanning. | Every two weeks for six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Marek, MD, Study Director — Molecular Neuroimaging / Institute for Neurodegenerative Disorders
Locations (1):
- Molecular Neuroimaging, LLC, New Haven, Connecticut, United States